CLINICAL TRIAL: NCT07380620
Title: Persistent Atrial Fibrillation in Southwest China Cohort Study-Stepwise Strategy for Treatment of Atrial Fibrillation Substrate Extended Study
Brief Title: Stepwise Strategy for Treatment of Atrial Fibrillation Substrate Extended Study
Acronym: SAFE-extended
Status: Enrolling by invitation | Type: Observational
Sponsor: Yuehui Yin (Other)
Responsible Party: Sponsor-Investigator, Yuehui Yin, MD, The Second Affiliated Hospital of Chongqing Medical University
Organization: The Second Affiliated Hospital of Chongqing Medical University (Other)
Other Study IDs: SAFE-extended study
Record Dates: First submitted 2025-09-28; First posted 2026-02-02 (Actual); Last update posted 2026-02-02 (Actual); Status verified 2026-01

CONDITIONS: Atrial Fibrillation
Keywords: Atrial Fibrillation
MeSH Terms: conditions — Atrial Fibrillation

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (6):
- normal LA group: the patients in this group have a normal size of left atrium.
- enlarged LA group: the patients in this group have an enlarged size of left atrium.
  Interventions: Other: other
- with HF group: the patients in this group suffer from heart failure.
  Interventions: Other: other
- without HF group: the patients in this group don't suffer from heart failure.
- HR control group: the patients in this group accept the therapy focus on heart rate control.
- Rhythm control group: the patients in this group accept the therapy focus on rhythm control.
  Interventions: Other: other

INTERVENTIONS:
Other: other — This study mainly describe the evolution and characteristic of patients with atrial fibrillation under different treatment plans and comorbidities.
  Groups: Rhythm control group; enlarged LA group; with HF group

SUMMARY:
This is an observational, bidirectional cohort study, aiming to establish a long-term registry of adult patients with Persistent atrial fibrillation (ps-AF) in Southwest China to characterize patient profiles and evaluate embolism risk, rate control, rhythm control and complication management and outcomes over 5 years' follow-up. The objectives of the study are to: Describe the demographic, clinical, and treatment characteristics of ps-AF patients across Southwest China and assess the effectiveness and safety of various AF treatment strategies, including oral anticoagulation, electrical cardioversion, catheter ablation, and left atrial appendage closure, in routine clinical practice. Identify patient- and treatment-related factors that influence therapeutic outcomes. Explore the characteristics of imaging multi-omics and blood multi-omics during follow-up. Explore the role of advanced technologies and artificial intelligence in improving procedural performance, risk stratification, and clinical decision-making in AF care. Participants will undergo standardized baseline evaluation and longitudinal follow-up to collect data on heart rhythm monitoring, treatment exposures, healthcare utilization, clinical events, and patient-reported outcomes. This cohort will generate real-world evidence to inform personalized and evidence-based management of AF.

DETAILED DESCRIPTION:
Background: Atrial fibrillation (AF) is estimated to affect over 33 million people worldwide and is associated with significant comorbidity such as embolism stroke, heart failure, dementia, etc. Consequently, AF poses a significant burden to the healthcare system, in both direct and indirect costs. The management of AF is complex, especially for patients with persistent AF, which is defined as sustained AF for > 7 days. It is preferable to terminate the AF and restore normal sinus rhythm for relief of symptoms associated with AF or improvement of cardiac structure and function. The maintenance of AF, especially persist AF is associated with fibrosis of left atria. Furthermore, AF itself promotes fibrosis, which in turn leads to increased conduction heterogeneity within the atrial substrate resulting in further progression of AF. In humans, atrial dilatation and degenerative changes have been observed. Persistent atrial fibrillation (AF) is a sustained form of AF associated with higher risks of stroke, heart failure, and mortality compared to paroxysmal AF. Managing persistent AF is challenging due to its complex mechanisms, lower success rates with standard treatments, and greater likelihood of recurrence. Research focuses on understanding its progression, identifying risk factors, and optimizing treatment strategies. Patients with persistent AF at diagnosis may differ in age, heart failure prevalence, and ejection fraction, but the pattern at diagnosis does not significantly affect ablation outcomes or AF recurrence rates.

Objectives: Describe the demographic, clinical, and treatment characteristics of ps-AF patients across Southwest China and assess the effectiveness and safety of various AF treatment strategies, including oral anticoagulation, electrical cardioversion, catheter ablation, and left atrial appendage closure, in routine clinical practice. Identify patient- and treatment-related factors that influence therapeutic outcomes. Explore the prevalence and treatment strategies of bradyarrhythmia in ps-AF patients. Explore the characteristics of imaging multi-omics and blood multi-omics during follow-up. Explore the role of advanced technologies and artificial intelligence in improving procedural performance, risk stratification, and clinical decision-making in AF care. Participants will undergo standardized baseline evaluation and longitudinal follow-up (prospective and retrospective) to collect data on heart rhythm monitoring, treatment exposures, healthcare utilization, clinical events, and patient-reported outcomes. This cohort will generate real-world evidence to inform personalized and evidence-based management of AF.

ELIGIBILITY:
Inclusion Criteria:

* Aged ≥18 years;
* diagnosed with persistent atrial fibrillation (ps-AF), defined as episodes lasting >7 days or requiring pharmacological/electrical cardioversion for rhythm restoration;
* Residing in Southwest China and capable of cooperating with long-term follow-up management;
* History of ps-AF treatment with complete medical records, and voluntary signing of the informed consent for long-term follow-up.

Exclusion Criteria:

* Comorbid severe hepatic/renal dysfunction or malignant tumors;
* Estimated survival period <1 year.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: persistent atrial fibrillation
Sampling Method: Non-Probability Sample
Enrollment: 5000 (Estimated)
Dates: Start 2025-10-09 (Actual); Primary Completion 2035-10-09 (Estimated); Study Completion 2035-12-31 (Estimated)

PRIMARY OUTCOMES:
Composite endpoint of stroke, major bleeding, worsening and new-onset heart failure, all-cause mortality | 5 years
  Composite endpoint of stroke, major bleeding, worsening heart failure, new-onset heart failure, and all-cause mortality
Major bleeding events, perioperative complications and adverse drug reactions | 5 years
  Major bleeding events (e.g., intracranial hemorrhage, gastrointestinal bleeding); Perioperative complications (e.g., pericardial tamponade, thrombus formation, vascular complications); Adverse drug reactions (e.g., anticoagulant-induced thrombocytopenia, amiodarone-induced thyroid dysfunction, prolonged QT interval, bradyarrhythmia, pulmonary fibrosis, etc.).

SECONDARY OUTCOMES:
Incidence of MACCE, SSS, AF recurrence and embolism events | 5 years
  Incidence of MACCE (Major Adverse Cardiovascular and Cerebrovascular Events); Sinus rhythm maintenance rate, AF recurrence time, duration of persistent recurrence (assessed via 12-lead ECG + Holter, defined as atrial arrhythmia lasting ≥30 seconds); Incidence of stroke or systemic embolism events.

CONTACTS AND LOCATIONS:
Locations (1):
- the second affiliated hospital of CQMU, Chongqing, China

IPD SHARING:
Plan to Share IPD: No
Sharing such data without the patient's explicit authorization may violate their right to privacy and contravene the informed consent terms obtained in the study.